CLINICAL TRIAL: NCT06377566
Title: BV-AVD in Patients With Newly-Diagnosed, Early Stage, Bulky Hodgkin Lymphoma Using a PET-adapted and MTV-guided Approach
Brief Title: A Study of BV-AVD in People With Bulky Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-039
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Ann Arbor stage I or II; Brentuximab vedotin; Doxorubicin HCL; Vinblastine Sulfate; Dacarbazine; Pembrolizumab; Gemcitabine; Vinorelbine
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; pembrolizumab; Gemcitabine; Vinorelbine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, investigator-initiated, single-arm phase II trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BV-AVD (brentuximab vedotin, doxorubicin, vinblastine, dacarbazine) (Experimental): All patients will receive 2 cycles of brentuximab vedotin (BV) in combination with AVD chemotherapy (doxorubicin, vinblastine, dacarbazine). Prophylactic growth factor support will be mandated with each cycle. After 2 cycles of therapy, patients will undergo FDG-PET/CT scan (PET2). Patients with disease progression (Deauville 4 or 5) will be taken off study. Patients who achieve a PETnegative scan (Deauville score of ≤ 3) will receive 2 additional cycles of BV-AVD with no further therapy. In those with partial response or stable disease (Deauville score of 4 or 5), patients will be stratified by baseline metabolic tumor volume (bMTV) as bMTV-high (> 150 cm3 ) or bMTV-low (≤ 150 cm3 ) as measured on pre-treatment FDG-PET/CT. In the bMTV-low group, patients will receive an additional 2 cycles of BV-AVD in combination with radiation therapy.
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Vinorelbine; Diagnostic Test: FDG-PET/CT scan

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin will be administered at 1.2 mg/kg IV on days 1 and 15 of each 28-day cycle
Drug: Doxorubicin — Doxorubicin 25 mg/m^2 IV
Drug: Vinblastine — Vinblastine 6 mg/m^2 IV
Drug: Dacarbazine — Dacarbazine 375 mg/m^2 IV on days 1 and 15 of each 28-day cycle
Drug: Pembrolizumab — Pembrolizumab will be administered at 200 mg IV (flat) on day 1
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 IV (days 1 an
Drug: Vinorelbine — Vinblastine 6 mg/m^2 IV
Diagnostic Test: FDG-PET/CT scan — After 2 cycles of therapy, patients will undergo FDG-PET/CT scan

SUMMARY:
The purpose of this study is to test whether BV-AVD is an effective treatment in people with early stage, bulky Hodgkin lymphoma that was recently diagnosed and who have not yet received any treatments for their disease.

BV is a type of drug called an antibody-drug conjugate (ADC). ADCs are a substance made up of a monoclonal antibody chemically linked to a drug. Antibodies are proteins made by the immune system to fight infections and other possible harms to the body. The monoclonal antibody binds to specific proteins or receptors found on certain types of cells, including cancer cells. The linked drug enters these cells and kills them without harming other cells. Researchers think BV may be an effective treatment for this type of cancer because the drug targets cells that have CD30, which play a role in cancer cell growth. By destroying these cells, BV may help slow or stop the growth of the cancer. AVD (doxorubicin, vinblastine, and dacarbazine) is a treatment regimen that works by stopping the growth of cancer cells, either by killing the cells or by stopping them from dividing. The researchers think that BV in combination with AVD may work better than AVD alone to slow or stop the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of classical, CD30-positive Hodgkin lymphoma confirmed at enrolling institution.
* Ann Arbor stage I or II FDG-avid disease by FDG-PET/CT.
* Disease bulk defined as any lymph node mass with transverse maximal diameter ≥ 7.0 cm or coronal maximal diameter ≥ 7.0 cm on CT imaging.
* Age 18 and over.
* ECOG Performance Status ≤ 2
* Females of childbearing age must be on an acceptable form of birth control per institutional standards during the treatment period.
* Males must consistently use an acceptable form of contraception per institutional standards during the treatment period.

Exclusion Criteria:

* Prior systemic therapy or radiation therapy for Hodgkin lymphoma (excluding corticosteroids)
* Cardiac ejection fraction < 50% as measured by echocardiogram.
* Platelet count ≤ 75,000/µL.
* Hemoglobin level ≤ 7.0 mg/dL.
* Absolute neutrophil count ≤ 1.0 K/µL.
* Serum creatinine clearance < 30 mL/minute as estimated by the Cockcroft-Gault Method.
* Transaminase levels > 3 times the upper limit of normal in the absence of a history of Gilbert's disease or hepatic involvement. In patients with Gilbert's disease, > 5 times the upper limit of normal is exclusionary.
* Total bilirubin ≥ 1.5 the upper limit of normal in the absence of a history of Gilbert's disease or hepatic involvement. In patients with Gilbert's disease, > 3 times the upper limit of normal is exclusionary.
* Pre-existing peripheral neuropathy ≥ grade 2 prior to participation.
* Known pregnancy or breast-feeding
* Active viral infection with hepatitis B or hepatitis C. For hepatitis B, patients who are seropositive (hepatitis B core Ab positive) are permitted if HBV DNA is negative by PCR. For hepatitis C, patients who are seropositive (hepatits C Ab positive) are eligible if HCV DNA is negative by PCR and curative therapy has been completed.
* Concurrent malignancy requiring active therapy within the last 2 years with the exception of basal cell or squamous cell carcinoma limited to the skin, carcinoma in situ of the cervix, breast or localized prostate cancer. Adjuvant hormonal therapy for cancer previously treated for curative intent is permitted.
* Patients with autoimmune conditions requiring active, ongoing systemic immunosuppressive therapy.
* Medical illness unrelated to Hodgkin lymphoma which in the opinion of the treating physician and/or principal investigator makes participation inappropriate.

Note: Patients with HIV infection are permitted to enroll but are required to be on antiretroviral regimens that are in accordance with the current International AIDS Society guidelines concurrently with chemotherapy. Use of experimental antiretroviral agents or those containing zidovudine or ritonavir, cobicistat or similar potent CYP3 inhibitors are prohibited. In order to be eligible, patients taking zidovudine or ritonavir, or cobicistat or other CYP3 inhibitors must change to a different regimen 7 days prior to therapy initiation. Subjects must be on HAART for at least 12 weeks prior to therapy.

Note: Patients with pre-existing autoimmune conditions are NOT excluded unless there is an autoimmune condition requiring active, ongoing systemic immunosuppressive therapy. However, careful consideration should be given to patients with pre-existing autoimmune conditions who may need pembrolizumab. Any concerns regarding patients with pre-existing autoimmune conditions and eligibility should be reviewed with the study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stuver, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm